CLINICAL TRIAL: NCT06928896
Title: Friction or Frictionless: What is the Most Effective Method for Retracting Anterior Teeth?
Acronym: Lam Le Nguyên
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Assoc.Prof.Dr. Nguyen Ngoc Rang, Faculty Odonto-Stomatology, Can Tho University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Le nguyên lâm ctump
Record Dates: First submitted 2024-10-15; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-10

CONDITIONS: Angle Class I; Alveolar Bone Loss
Keywords: alveolar bone, elastomeric chains, friction, frictionless
MeSH Terms: conditions — Malocclusion, Angle Class I; Alveolar Bone Loss | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1. Using the friction (Experimental)
  Interventions: Procedure: This interventional trial enrolled a total of 42 patients, dividing them into two age groups: group 1. Using the friction and group 2. Using the frictionless
- Group 2. Using the frictionless (Experimental)
  Interventions: Procedure: This interventional trial enrolled a total of 42 patients, dividing them into two age groups: group 1. Using the friction and group 2. Using the frictionless

INTERVENTIONS:
Procedure: This interventional trial enrolled a total of 42 patients, dividing them into two age groups: group 1. Using the friction and group 2. Using the frictionless — Cone beam computed tomography (CBCT) was conducted before and after retraction to evaluate alveolar changes and speed.

SUMMARY:
Objective:To evaluate the effectiveness of the friction (sliding mechanism with elastomeric chains) and frictionless (T-loop) methods for retracting anterior teeth in Angle Class I malocclusion.

Methods: This clinical intervention study examined the duration of maxillary incisor retraction from August 2022 to August 2024 in 42 adult patients who had completed canine retraction. The process involved resolving horizontal and vertical discrepancies, establishing a Class I relationship between the canines, and altering the overbite (the interproximal space between the lateral incisors and canines) until an ideal overbite index of 2 mm was achieved. Cone beam computed tomography (CBCT) was conducted before and after retraction to evaluate alveolar changes and speed.

DETAILED DESCRIPTION:
Step 1. The following data were collected: general information, clinical examination, classification of facial symmetry while facing forward, profile, state of the temporomandibular joint, relationships between the first molar teeth, and canine relationship. Patients with bilateral type I angle malocclusion were selected. The PAR(W) index was calculated using the model cast as a measurement. Subsequently, the patients' model casts, standardized intraoral and extraoral photographs, panoramic films, and cephalometric films were used to make the second selection. A patient's upper first premolar was removed if orthodontic treatment was indicated. All cephalometric films that met the study's requirements were analyzed using the customized software WebCeph. Before beginning orthodontic therapy, the bleeding time, clotting time, and platelet count were tested in the patients who met the inclusion criteria. Before participating in the study, patients signed a permission form and received information about the study's goals and methods.

Step 2. The TransbondTM XT Light Cure Adhesive and the Victory Series Metal Bracket System (MBT 0.022 slot, 3M Unitek®, USA) were employed. This study used a two-step space closure method for tooth extraction, in which the canine is moved backward to obtain a Class I canine relationship, and the relationship between the molars is changed if necessary. Subsequently, CTCB was performed before the procedure of retracting the four incisors. At this stage, the patient's group allocation was determined randomly. IZC mini-screws (8 x 1.6 mm, 3M UnitekTAD, St. Paul, Minn.) were used in both groups .

In group 1 (sliding mechanism: using elastomeric chains combined with mini-screws), 3M elastomeric chains were used to retract the four maxillary incisors toward the mini-screws with 160 g of force.

In group 2 (loop mechanism), the T-loop was measured and bent using TMA wire (0.016 × 0.022 inches, 3M, USA) to conform to the patient's arch. The loop was positioned distal to the lateral incisor to initiate the force and modify the loop. Weingart forceps were utilized to retract the archwire posterior to the first premolar, expanding the loop by about 4 mm (150 g) and securing the tail to initiate activation. The loop force was adjusted to fully close space at each subsequent visit. To enhance anchoring, the mini-screw was placed identically on both sides of the arch (the screw positioning resembled that of group 1). Subsequently, the upper first molar was secured to the mini-screws using a 0.012-inch diameter ligature wire.

After the retraction of four incisors, post-retraction CBCT scans were obtained, and the retraction of the four upper incisors was analyzed (overbite achieved 2 mm, Class I canine relationship). CBCT images were generated in DICOM format and imported into Ondemand3Ddental software (Cybermed, Korea, version 1.0.11.1007) for data measurement. The teeth were identified using axial navigation guidance from the multi-planar reconstruction (axial, sagittal, and coronal) of the CBCT, following the measurement method in Le's study (2023) , while ensuring that radiation exposure was kept as low as reasonably achievable (ALARA Guidelines)

ELIGIBILITY:
Inclusion Criteria:

* Angle class I malocclusion on one or both sides
* Without any previous orthodontic treatment
* Indications for fixed appliances, premolar extraction to create space during treatment
* Consented to participate in the study

Exclusion Criteria:

* History of craniofacial traumas, anomalies, congenital defects, or systemic diseases related to osteogenic metabolisms, e.g. diabetes mellitus, kidney diseases, osseous diseases
* Patients took anticoagulant drugs that affected bone metabolism (eg., for example, heparin, warfarin, NSAIDs, cyclosporine, glucocorticoids, medroxyprogesterone acetate, etc.)
* Mini screw, and hook failure

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of the friction (sliding mechanism with elastomeric chains) and frictionless (T-loop) methods for retracting anterior teeth in Angle Class I malocclusion. | 6 months after enrollment
  This interventional trial enrolled a total of 42 patients, dividing them into two age groups: group 1. Using the friction (sliding mechanism-elastomeric chains) and group 2. Using the frictionless (T-loop). For each patient, cone beam computed tomography (CBCT) was taken before and after retraction to evaluate alveolar changes.
  Study variables measured on CBCT. The palatal plane (PP) represents the magnetic connection between the PNS (posterior nasal spine) and the ANS (anterior nasal spine), V: a vertical reference line perpendicular to the ANS-PNS line, H: a vertical reference line parallel to the ANS-PNS line. Four lines perpendicular to the V line (L0, L1, L2, L3, 2 mm apart). Line L0 passes through the cementoenamel junction (CEJ) on the buccal side. Measure the alveolar bone thickness at 3 positions (S1, S2, S3, lingual, and buccal) at T1 and T2.

CONTACTS AND LOCATIONS:
Locations (1):
- Can Tho University of Medicine and Pharmacy, Can Tho, Can Tho City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vazquez E. Saquinavir plus ritonavir reduce viral load by 99.9 percent. Posit Aware. 1996 Nov-Dec;7(6):8-9. PMID 11363983
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39230024/